CLINICAL TRIAL: NCT03060811
Title: Mediterranean Diet, Trimethylamine N-oxide (TMAO) and Anti-oxidants in Healthy Adults
Acronym: TMED
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Prof. Silvia Savastano, Researcher/Adjunct Professor, Federico II University
Other Study IDs: 173/16
Record Dates: First submitted 2017-02-14; First posted 2017-02-23 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Mediterranean Diet; Trimethylamine N-oxide; Cardiovascular Risk Factor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Trimethylamine N-oxide (TMAO) is a small organic compound naturally present in fish and seefood or generated by the bacterial breakdown of dietary phosphatidylcholine and carnitine-containing foods within the human gut microbiome. Elevated serum TMAO was previously reported to be associated with an elevated risk for cardiovascular events.

Aim of this study was to investigate the association between plasma levels of TMAO with the Mediterranean diet in a cohort of healthy adults.

ELIGIBILITY:
Inclusion Criteria:

healthy subjects of both gender

Exclusion Criteria:

* age>65 years
* > BMI 30 kg/m2
* vegetarians
* smokers
* gastrointestinal diseases or complaints
* chronic illnesses or other metabolic diseases (including trimethylaminuria)
* abnormal blood chemistry values indicative of organ dysfunctions
* nutritional supplements, antibiotics or probiotics within 2 months of recruitment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects (n=84) aged 21-50 years with a BMI of 20-29.9 kg/m2, chosen among hospital volunteers and employees from the same geographical area. A sample size of n=40 was determined from a power analysis of a within-subject design to detect a 10% difference of plasma TMAO concentration at alfa<0.05 and β =0.8. Participants were screened by the use of a blood chemistry profile, cell count, and health history questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-09-22 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Adherence to Mediterranean Diet by Predimed Questionnaire | September 2016 to December 2016
  Validated 14-item tool of adherence to the Mediterranean diet, with three categories of adherence (≤5, low adherence, 6-9, average adherence and ≥10 points, high adherence)
Trimethylamine N-oxide plasma levels | September 2016 to December 2016
  ultra high-performance liquid chromatography

SECONDARY OUTCOMES:
cardiovascular risk | September 2016 to December 2016
  metabolic syndrome parameters; Homa Index; Framingham score; ASCVD Risk Estimator

IPD SHARING:
Plan to Share IPD: No